CLINICAL TRIAL: NCT03907046
Title: Anticoagulation in Intracerebral Hemorrhage (ICH) Survivors for Stroke Prevention and Recovery
Brief Title: Anticoagulation in ICH Survivors for Stroke Prevention and Recovery
Acronym: ASPIRE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2000026409; 1U01NS106513-01A1 (NIH)
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Intracerebral Hemorrhage; Atrial Fibrillation
MeSH Terms: conditions — Cerebral Hemorrhage; Atrial Fibrillation | interventions — apixaban; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Apixaban (Active Comparator): Apixaban dosing will be 5 mg tablet in morning and 5 mg tablet in evening. A reduced dose of 2.5 mg tablet in morning and 2.5 mg tablet in evening will be used if: (1) ≥2 of the following are present: age ≥80 years, body weight ≤60 kg, or serum creatinine 1.5-2.4 mg/dL, or (2) Patient is taking a strong CYP3A4/pGP inhibitor (e.g., ketoconazole, itraconazole, ritonavir, or clarithromycin).
  Interventions: Drug: Apixaban
- Aspirin (Placebo Comparator): Aspirin dose will be 81 mg tablet once daily.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Apixaban — Apixaban is an oral anticoagulant of the Factor Xa inhibitor class.
  Other Names: Eliquis
  Arms: Apixaban
Drug: Aspirin — Aspirin is an oral antiplatelet drug.
  Arms: Aspirin

SUMMARY:
Primary Aim: To determine if apixaban is superior to aspirin for prevention of the composite outcome of any stroke (hemorrhagic or ischemic) or death from any cause in patients with recent ICH and atrial fibrillation (AF).

Secondary Aim: To determine if apixaban, compared with aspirin, results in better functional outcomes as measured by the modified Rankin Scale.

DETAILED DESCRIPTION:
ASPIRE is a randomized, double-blinded, phase III clinical trial designed to test the efficacy and safety of anticoagulation, compared with aspirin, in patients with a recent ICH and non-valvular AF. Seven hundred patients will be enrolled over 3.5 years and followed for study outcomes for a minimum of 12 months and maximum of 36 months. The primary efficacy outcome is any stroke (hemorrhagic or ischemic) or death from any cause. The secondary efficacy outcome is the change in the modified Rankin Scale score. Recruitment will take place at sites coordinated through the NIH/NINDS StrokeNet.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Intracerebral hemorrhage (ICH) (including primary intraventricular hemorrhage) confirmed by brain CT or MRI
* Can be randomized within 14-180 days after ICH onset
* Non-valvular AF (defined as atrial fibrillation or atrial flutter), documented by electrocardiography or a physician-confirmed history of prior AF
* Provision of signed and dated informed consent form by patient or legally authorized representative
* For females of reproductive potential: use of highly effective contraception

Exclusion Criteria:

* Index event is hemorrhagic transformation of a brain infarction or hemorrhage into a tumor
* History of earlier ICH within 12 months preceding index event
* Active infective endocarditis
* Clear indication for anticoagulant drugs (e.g., requires anticoagulation for deep vein thrombosis or pulmonary embolism) or antiplatelet drugs (e.g., requires aspirin or clopidogrel for recent coronary stent).
* Previous or planned left atrial appendage closure
* Clinically significant bleeding diathesis
* Serum creatinine ≥2.5 mg/dL
* Active hepatitis or hepatic insufficiency with Child-Pugh score B or C
* Anemia (hemoglobin <8 g/dL) or thrombocytopenia (<100 x 10^9/L) that is chronic in the judgment of the investigator
* Pregnant or breastfeeding
* Known allergy to aspirin or apixaban
* Concomitant participation in a competing trial
* Considered by the investigator to have a condition that precludes safe or active participation in the trial
* Persistent, uncontrolled systolic blood pressure (≥180 mm Hg)
* ICH caused by an arteriovenous malformation (AVM) that has not yet been secured

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Stroke or death | Up to 3 years
  Incidence of stroke of any type (ischemic or hemorrhagic) or death from any cause

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) score | Change from baseline to 12 months; change over duration of follow-up
  Measure of neurologic disability (0=no disability to 6=dead)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin N Sheth, MD, Principal Investigator — Yale University; Hooman Kamel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (183):
- United States (183):
  - University of Alabama Hospital, Birmingham, Alabama
  - University of South Alabama University Hospital, Mobile, Alabama
  - Chandler Regional Medical Center, Chandler, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - UAMS Medical Center, Little Rock, Arkansas
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Medical Center, Castro Valley, Castro Valley, California
  - Arrowhead Regional Medical Center, Colton, California
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Kaiser Permanente Fontana Medical Center, Fontana, California
  - Community Regional Medical Center of Fresno, Fresno, California
  - St. Jude Medical Center, Fullerton, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Los Alamitos Medical Center, Los Alamitos, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Doctors Medical Center Modesto, Modesto, CA, Modesto, California
  - Hoag Hospital Newport Beach, Newport Beach, California
  - UC Irvine Medical Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Huntington Memorial Hospital, Pasadena, California
  - Kaiser Permanente Redwood City Medical Center, Redwood City, CA, Redwood City, California
  - UC Davis Medical Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - San Francisco General Hospital, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Stanford University Medical Center, Stanford, California
  - PIH Health Hospital - Whittier, Whittier, California
  - University of Colorado Hospital, Aurora, Colorado
  - St. Mary's Medical Center, Grand Junction, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - New Hanover Regional Medical Center, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Ascension Sacred Heart Pensacola, Pensacola, Florida
  - Cleveland Clinic Tradition Hospital, Port Saint Lucie, Florida
  - Tampa General Hospital, Tampa, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Regional Medical Center - Boise, Boise, Idaho
  - NCH Hospital, Arlington Heights, Arlington Heights, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Javon Bea Hospital - Riverside, Rockford, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - University of Iowa Medical Center, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Ochsner Medical Center - Main Campus, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Flint, Flint, Michigan
  - Trinity Health Saint Mary's, Grand Rapids, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - HealthPartners Methodist Hospital, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, St. Paul, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Health Care, Columbia, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Cox Medical Center South, Springfield, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Capital Health Regional Medical Center, Trenton, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Kings County Hospital Center, Brooklyn, New York
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - NYC Health + Hospitals/Elmhurst, Elmhurst, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai West, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - NYP Columbia University Medical Center, New York, New York
  - NYP Weill Cornell Medical Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Strong Memorial Hospital, Rochester, New York
  - Staten Island University Hospital - North Campus, Staten Island, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Burke Rehabilitation Center, White Plains, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - ECU Health Medical Center, Greenville, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - UH Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - OU Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Ascension St. John Medical Center, Tulsa, Oklahoma
  - St. John Medical Center, Tulsa, Oklahoma
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - PeaceHealth Sacred Heart Medical Center - RiverBend, Springfield, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina University Hospital, Charleston, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Erlanger Health System, Chattanooga, Tennessee
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - Semmes Murphey Main Campus, Memphis, Tennessee
  - Vanderbilt University Hospital, Nashville, Tennessee
  - St. David's Medical Center, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - The University of Vermont Medical Center, Burlington, Vermont
  - UVA Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Medical Center - Cherry Hill Campus, Seattle, Washington
  - WVU Healthcare Ruby Memorial Hospital, Morgantown, West Virginia
  - Froedtert Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520